CLINICAL TRIAL: NCT04361435
Title: Comparison of Two Methods to Airway Clearance in Patients Admitted to Intensive Care Unit for COVID-19: A Pilot Corssover Randomized Controlled Trial
Brief Title: Lung Recruitment Device for COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Dymedso Inc. (Unknown); Réseau de Recherche en Santé Respiratoire du Québec (Unknown); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Philippe Jouvet, Professor, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-21-2020-2871
Record Dates: First submitted 2020-04-12; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Physiotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of the 2 arms (None-invasive oscillating device (NIOD) first or chest physiotherapy (CPT) first). Random allocation will be generated by an independent investigator in an equal number assigned to each intervention. Stratification will be applied for age (>18 years or =<18 years of age) and sites (CHUSJ and General Hospital).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIOD first (Other): In this arm, we will apply for NIOD first which will be performed by non-physiotherapists such as respiratory therapists and bedside nurses. This arm of patients will receive standard CPT at least 3 hours after the NIOD intervention.
  Interventions: Procedure: Chest physiotherapy using a non-invasive oscillating device
- CPT first (Other): In this arm, we will apply for CPT first which will be performed by physiotherapists. This arm of patients will receive NIOD procedures which will be performed by non-physiotherapists such as respiratory therapists and bedside nurses at least 3 hours after the CPT intervention.
  Interventions: Procedure: Chest physiotherapy using a non-invasive oscillating device

INTERVENTIONS:
Procedure: Chest physiotherapy using a non-invasive oscillating device — NIOD will be implemented on four different parts of the chest walls, 3 minutes for each part and 12 minutes in total per each session. Left and right front and posterior chest walls will be stimulated, particularly, on the anterior chest, intercostal spaces 1-2 above nipple line and lateral side of the mid-clavicular line 1-2 below intercostal spaces. The intensity of the NIOD can be selected between 80-100%, which is pre-specified on the machine.

SUMMARY:
INTRODUCTION As there is no specific cure in the treatment of COVID-19 at this moment of the pandemic, supportive management including mechanical ventilation is the core management in an intensive care unit (ICU). It is a challenge to provide consistent care in this situation of high demand and potential staff shortage in ICU. Also, the investigators need to reduce unnecessary exposure of the providers to the virus. This study aims to examine the impact of care using a non-invasive oscillating device (NIOD) for chest physiotherapy in the care of mechanically ventilated patients with COVID-19.

METHODS Objective: To explore if a NIOD performed by non-specialized personnel is not inferior to the standard Chest PhysioTherapy (CPT) in the care of COVID-19.

Design: A Pilot Multicenter Prospective Crossover Randomized Study. Setting: Two ICUs in Canadian Academic Hospitals (CHU Sainte Justine and Montreal General Hospital) Patients: All the mechanically ventilated patients admitted to the two ICUs, and CPT ordered by the responsible physician, with COVID-19 infection during the study period.

Procedure: The investigators will implement NIOD and CPT alternatingly for 3 hours apart over 3 hours. We will apply a pragmatic design, so that other procedures including hypertonic saline nebulization, Intermittent Positive Pressure Ventilation (IPPV), suctioning (e.g., oral or nasal), or changing the ventilator settings or modality can be provided at the direction of bedside intensivists in charge. The order of the procedures (i.e. NIOD or CPT) will be randomly allocated.

Measurements and Analyses: The primary outcome measure is the oxygenation level before and after the procedure (SpO2/FIO2 (SF) ratio). For the cases with Invasive ventilation and non-invasive ventilation, the investigators will also document expiratory tidal volume, vital signs, and any related complications such as vomiting, desaturations, or unexpected extubations. The investigators will collect the data before, 10 minutes after, and 30 minutes after the procedure.

Sample Size: The investigators estimate the necessary sample size as 25 for each arm (Total 50 cases), with a power of 0.90, alfa of 0.05, with the non-inferiority design.

FUTURE CONSIDERATIONS This randomized pilot study will be considered a running phase if the investigators can/should undertake the RCT which should follow without significant modification of the methods.

DETAILED DESCRIPTION:
1. BACKGROUND During COVID-19 pandemic, although the proportion of severe or fatal cases may vary by location, 15-30% of hospitalized patients were admitted to the intensive care unit in Italy and China (1-4).

   Pneumonia appears to be the most frequent serious manifestation of infection. In addition to respiratory symptoms, gastrointestinal symptoms have also been reported (2, 3, 5). The symptomatic infection can range from mild to critical; but, generally, the clinical course seems to have characteristics of slow progression from upper airway to the lower and the other systemic organs such as cardiac muscles. Radiographic findings include ground-glass opacities, crazy paving appearance, air space consolidation, broncho-vascular thickening in the lesion with a slow progression up until 10-14 days from the onset of disease (6-8).

   Staff Shortage & Protection Protecting the workforce is another critical challenge. Sick leaves or self-isolation has increased already. Caring for infected patients represents a substantial exposure risk for ICU staffs because of high and prolonged exposure to critically ill patients who presumably have higher viral shedding. This should be particularly noted for physiotherapists to whom chest physiotherapy can be prescribed more often than usual in this situation of ICU demand. On the other hand, only a limited number of physiotherapists are available in most of ICUs.

   Airway obstruction due to the production of secretion particularly with respiratory muscle weakness in critically ill is a major problem in clinical management. CPT has been proposed to assist in the clearance of tracheobronchial secretions. Techniques such as the conventional CPT with chest percussion and vibration, chest shaking and directed coughing may help to mobilize secretions towards the trachea and trigger coughing that could help to remove the secretions. However, a recent systematic review reported that there is no sufficient evidence to provide CPT in routine practice with a significant heterogeneity of the procedure techniques used (9-13).

   Extra-thoracic non-invasive oscillating devices (NIOD) are designed to interrupt the expiratory airflow and can help to secretions clearance. NIOD requires less patient cooperation and could be used without interruptions such as due to coughing or suctioning of secretion. Frequencer® (Dymedso, Montreal Canada) is a NIOD that locally target the affected lung areas. The safety has been attested particularly in patients with cystic fibrosis. In addition, this NIOD can be easily administered by non-specialized personnel such as respiratory therapists or registered nurses (14, 15).

   This proposed study is to compare the effectiveness of NIOD performed by non-specialized personnel (respiratory therapist, nurse, physicians) versus standard CPT performed by a physiotherapist.
2. OBJECTIVES & RESEARCH QUESTIONS Objectives

This project has 3 specific objectives:

1. To study the feasibility and tolerance of NIOD in the mechanically ventilated patients
2. To study if NIOD performed by non-specialized personnel is not inferior to the standard CPT done by the physiotherapist in the care of COVID-19.
3. To study the impact of NIOD and CPT on oxygenation. Research questions to be asked

1. Is the NIOD safe and well-tolerated to be applied to critically ill patients with COVID-19? 2. Is the NIOD not inferior to standard CPT performed by a physiotherapist with respect to the effect of oxygenation in critically ill COVID-19 patients? 3. What kinds of physiological positive effects can the NIOD and CPT provide on critically ill patients with COVID-19? 3. SIGNIFICANCE This study will provide valuable knowledge about secretion management in critically ill patients. It will also contribute to more efficient health care practice and resource utilization (i.e., physiotherapist).

To be specific, NIOD could improve the respiratory management of patients with COVID-19. The findings acquired in this study can be generalizable to other hospitals and cohorts in ICUs. Ultimately, this could reduce the impact of COVID-19 on the health system and could reduce the exposure of physiotherapists to COVID-19.

4. METHODS 4.1 Study Design The investigators will adopt a prospective crossover non-inferiority randomized design.

4.2 Setting Two ICUs in CHU Sainte Justine (Pediatric ICU) and Montreal General (Adult ICU) Hospital.

4.3 Screening of Eligible Patients and Informed Consent Procedure. When there is a potentially eligible patient, a research assistant will be notified in 24/7 during the study period. The investigators will obtain the informed consent (IC) from patients or parents/guardians using an informed consent form.

4.4 Eligible Patients Please see the other section of this application. 4.5 Intervention: Each subject will receive the NIOD (i.e., Frequencer) and the standardized CPT for this study.

4.5.1 Suctioning and Other Interventions As per each ICU's protocol, the participants will have a suction of secretion as needed. Any other potential interventions such as nebulization of hypertonic saline and bronchodilator and that with a metered-dose inhaler (MDI) can be given without any restrictions.

4.5.2 Positioning All the procedures (i.e., NIOD and CPT) will be applied with any positioning such as sitting and prone positions. Caregivers can also change the positioning as needed during the procedures. All the outcome parameters should be measured (before and after the procedures) with the same positioning.

4.5.3 Detailed Procedure NIOD will be implemented on four different parts of the chest walls, 3 minutes for each part and 12 minutes in total per each session. Left and right front and posterior chest walls will be stimulated, particularly, on the anterior chest, intercostal spaces 1-2 above nipple line and lateral side of the mid-clavicular line 1-2 below intercostal spaces. The intensity of the NIOD can be selected between 80-100%, which is pre-specified on the machine. The step-by-step procedure is described in the Appendix.

4.5.4 Selection of the Membrane There are several selections of the membrane available. The investigators will use the membrane according to the manual provided by the manufacture.

4.5.5 Standardization of the Procedure. The procedure using the NIOD will be standardized. The investigators will use a video clip (i.e., YouTube) and will ask each caregiver to view at least once before the first procedure of the day.

4.5.6 CPT. CPT will be defined as an assistant strike to the chest wall repeatedly with a cupped hand in specific places. CPT will be performed by a physiotherapist as per protocol in each institution.

4.6 Detailed Protocol Patients satisfying the eligibility criteria will have their baseline data collected prior to the intervention.

Randomization Participants will be randomized into one of the 2 arms (NIOD first or CPT first). In the existing studies targeting adults, 20-60Hz are most widely used (personal communication with Dymedso Inc.). The investigators will apply 40Hz. Randomization will be carried out by the independent research assistant in CHU Sainte Justine (CHUSJ). Random allocation will be generated by an independent investigator in an equal number assigned to each intervention. Stratification will be applied for age (>18 years or =<18 years of age) and sites (CHUSJ and General Hospital) (Figure2).

Timing of the Data Measurement The data measured in mechanical ventilation and patients monitor will be collected 1) right before the intervention being initiated, 2) 10 minutes after the end of the intervention, and 3) 30 min after each intervention finished. The investigators will manually record the following variables for the three timings (4.9.1). Vital sign values including EtCO2 waveforms from the beginning of the intervention until 30 min after the intervention will be extracted from the Electronic Medical Records (i.e., every minute) for the cohorts in CHUSJ.

4.7 Sample Size Calculation A trial aims to determine whether NIOD will be able to provide an improvement of oxygenation not inferior to standard CPT. The investigators estimate the mean improvement of SF ratio is 30 with a variance of 10 in CPT. It was claimed to be clinically non-inferior if effect of NIOD was 20% lower than the standard CPT. The largest clinically acceptable difference of 6 (30*0.20) is declared that NIOD is non-inferior compares with CPT. Type I, II error and ratio are set at 0.05, 0.1, and 1:1. With this, we require 32 cases in total (16 cases per group). Considering this, we will collect 25 cases per group (16-21).

4.8 Protocol Violation. Protocol violation in eligibility is defined as when a patient was randomized but does not follow the protocol. These patients will be excluded from the analyses. Patients who withdraw their consent after randomization will be excluded from the analyses. The number of excluded patients after randomization will be displayed in the CONSORT flow diagram (Fig3). Patients assigned to both arm receive the standard ICU care in each center.

4.9 Statistical Analyses The main analysis will be performed according to the intention-to-treat (ITT) principle. A patient who withdrew consent or patients with a protocol violation concerning eligibility are excluded from ITT analyses. Differences in patient characteristics between patients lost to follow-up and included patients will be assessed. In view of the non-inferiority study design, per-protocol (PP) analyses will also be performed. All subjects from the ITT population without protocol violations and deviations regarding treatment will be included in the PP population. The investigators will also repeat the analyses with logistic regression to consider that randomization was stratified by the participating center and age (>18 or =<18 years of age). Non-inferiority will be established if the lower limit of the one-sided 95% confidence for the mean of SF ratio for CPT group relative to that of patients with NIOD exceeds the critical value corresponding to the absolute 5% margin below the observed proportion under usual care. All statistical analyses will be conducted with Stata (Stata Corp LP, TX USA) or other statistical software(s).

5. ETHICAL CONSIDERATIONS 5.1 Overview The device and membrane for adults applied have been certified and approved by Health Canada and commercially available in Canada (Fig1a). Although the prototype transducer for infants (Fig1b) has not been tested on patients as a large trial, the mechanism of the pressure delivery and the intensity of the delivering pressure/ oscillation should be similar as compared to the existing model for children and adult patients. The devices have been approved by Health Canada. The investigators believe there should be no excessive harm as compared to the current standard CPT. Patients will also receive standard CPT during the study period, which is widely accepted as a practice for airway clearance in the ICUs.

This study will be approved by the Health Research Ethics Board of the University of Montreal, Canada. The study protocol will be registered into https://clinicaltrials.gov/ once it is approved by the local IRB.

5.2 Risk Minimization and Data and Safety Monitoring Board (DSMB) It has shown that NIOD was feasible and well-tolerated in adult and relatively older children. For this study, another DSMB will be in place to independently supervise any potential side effects. It will include Francois Proulx MD and Tse Man Sze MD. The DSMB will follow the study completion and review any significant potential complications related to the intervention with NIOD. Any occurrence of pneumothorax, need for unplanned intubation, life-threatening event, during or in the 2 hours following the study, will be declared to and reviewed by the DSMB, which will independently decide on the need to stop or continue the study.

ELIGIBILITY:
All the patients admitted to the ICUs during the study period will be screened. We will not set any restrictions regarding the timing of the prescription of CPT (i.e., length of ICU stay before screening) for the screening. We will include only if CPT is expected to be used as management at least for the next 24 hours in the ICUs from the time of inclusion. For instance, if CPT will be expected to be discontinued from the management in a day, we will exclude them from the inclusion. CPT can be prescribed for airway clearance with any etiology such as atelectasis at the directions of bedside intensivists in charge of the study date.

Specific Inclusion criteria

* Patients diagnosed as COVID-19
* Patents strongly suspected its infection and the result of virological testing is pending as of screening.
* Patients with any type of mechanical ventilation (i.e., Invasive, non-invasive, high flow nasal therapy)
* Patients are on standard oxygen by mask or nasal cannula and the FiO2 provided can be measurable.
* Patients who are on respiratory monitoring at least SpO2 can be continuously measurable.

Exclusion Criteria:

* CPT order will (or is expected to) be discontinued within 12 hours from the inclusion timing. This may include potential discharge from the unit.
* CPT is not ordered for airway clearance.
* SpO2 is not stable (SpO2=<80%) with more than 0.60 of FIO2 for ventilated patients including patients on NIV, at least for the previous 1 hour from the screening.
* SpO2 is not stable (SpO2=<80%) with more than 0.60 of FIO2 for the patients on HFNC, at least for the previous 1 hour from the screening.
* Bradycardia (HR<50bpm) at any intervention at least 24 hours before the screening.
* Patients with known pneumothorax, osteomyelitis at ICU admission.
* Thoracotomy within 1 month from the admission date.
* Known recent/unhealed rib fractures.
* Known skin injury of the chest wall.
* No, obtain of IC.
* Brain death or vegetated states.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
SpO2/FIO2 Ratio | 10 minutes and 30 minutes from the end of the procedure
  Difference before the procedure and 10 minutes from the end of the procedure

SECONDARY OUTCOMES:
Blood pressures | 10 minutes and 30 minutes from the end of the procedure
  Changes in values
Heart rates | 10 minutes and 30 minutes from the end of the procedure
  Changes in values
Respiratory rate | 10 minutes and 30 minutes from the end of the procedure
  Changes in values
Body temperature | 10 minutes and 30 minutes from the end of the procedure
  Changes in values
Modified Wood Clinical Asthma Score (m-WCAS) | 10 minutes and 30 minutes from the end of the procedure
  Changes in values (0 to 10, worse outcome is 10)
Expiratory tidal lung volume. | 10 minutes and 30 minutes from the end of the procedure
  Changes in volume.
End-tidal CO2 | 10 minutes and 30 minutes from the end of the procedure
  Changes in values and blood gas parameters.
Clinical Respiratory severity scores. | 10 minutes and 30 minutes from the end of the procedure
  Changes in scores

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jouvet, MD PhD MBA, Principal Investigator — St. Justine's Hospital

IPD SHARING:
Plan to Share IPD: No
All the study documents will be shared only among the two sites. The summarized cleaned data will be shared with the co-investigators in both study sites.

REFERENCES:
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Kanne JP, Little BP, Chung JH, Elicker BM, Ketai LH. Essentials for Radiologists on COVID-19: An Update-Radiology Scientific Expert Panel. Radiology. 2020 Aug;296(2):E113-E114. doi: 10.1148/radiol.2020200527. Epub 2020 Feb 27. No abstract available. PMID 32105562
- [Result] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Result] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Result] Roque i Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2016 Feb 1;2(2):CD004873. doi: 10.1002/14651858.CD004873.pub5. PMID 26833493
- [Result] Chaves GS, Freitas DA, Santino TA, Nogueira PAM, Fregonezi GA, Mendonca KM. Chest physiotherapy for pneumonia in children. Cochrane Database Syst Rev. 2019 Jan 2;1(1):CD010277. doi: 10.1002/14651858.CD010277.pub3. PMID 30601584
- [Result] Hough JL, Flenady V, Johnston L, Woodgate PG. Chest physiotherapy for reducing respiratory morbidity in infants requiring ventilatory support. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD006445. doi: 10.1002/14651858.CD006445.pub2. PMID 18646156
- [Result] Lauwers E, Ides K, Van Hoorenbeeck K, Verhulst S. The effect of intrapulmonary percussive ventilation in pediatric patients: A systematic review. Pediatr Pulmonol. 2018 Nov;53(11):1463-1474. doi: 10.1002/ppul.24135. Epub 2018 Jul 18. PMID 30019451
- [Result] Ferreira LL, Valenti VE, Vanderlei LC. Chest physiotherapy on intracranial pressure of critically ill patients admitted to the intensive care unit: a systematic review. Rev Bras Ter Intensiva. 2013 Oct-Dec;25(4):327-33. doi: 10.5935/0103-507X.20130055. PMID 24553515
- [Result] Schieppati D, Germon R, Galli F, Rigamonti MG, Stucchi M, Boffito DC. Influence of frequency and amplitude on the mucus viscoelasticity of the novel mechano-acoustic Frequencer. Respir Med. 2019 Jul;153:52-59. doi: 10.1016/j.rmed.2019.04.011. Epub 2019 May 27. PMID 31163350
- [Result] Cantin AM, Bacon M, Berthiaume Y. Mechanical airway clearance using the frequencer electro-acoustical transducer in cystic fibrosis. Clin Invest Med. 2006 Jun;29(3):159-65. PMID 17058435
- [Result] Adams JY, Rogers AJ, Schuler A, Marelich GP, Fresco JM, Taylor SL, Riedl AW, Baker JM, Escobar GJ, Liu VX. Association Between Peripheral Blood Oxygen Saturation (SpO2)/Fraction of Inspired Oxygen (FiO2) Ratio Time at Risk and Hospital Mortality in Mechanically Ventilated Patients. Perm J. 2020;24:19.113. doi: 10.7812/TPP/19.113. Epub 2020 Jan 31. PMID 32069205
- [Result] Bilan N, Dastranji A, Ghalehgolab Behbahani A. Comparison of the spo2/fio2 ratio and the pao2/fio2 ratio in patients with acute lung injury or acute respiratory distress syndrome. J Cardiovasc Thorac Res. 2015;7(1):28-31. doi: 10.15171/jcvtr.2014.06. Epub 2015 Mar 29. PMID 25859313
- [Result] Ghazal S, Sauthier M, Brossier D, Bouachir W, Jouvet PA, Noumeir R. Using machine learning models to predict oxygen saturation following ventilator support adjustment in critically ill children: A single center pilot study. PLoS One. 2019 Feb 20;14(2):e0198921. doi: 10.1371/journal.pone.0198921. eCollection 2019. PMID 30785881
- [Result] Koyauchi T, Yasui H, Enomoto N, Hasegawa H, Hozumi H, Suzuki Y, Karayama M, Furuhashi K, Fujisawa T, Nakamura Y, Inui N, Yokomura K, Suda T. Pulse oximetric saturation to fraction of inspired oxygen (SpO2/FIO2) ratio 24 hours after high-flow nasal cannula (HFNC) initiation is a good predictor of HFNC therapy in patients with acute exacerbation of interstitial lung disease. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620906327. doi: 10.1177/1753466620906327. PMID 32046604
- [Result] Kwack WG, Lee DS, Min H, Choi YY, Yun M, Kim Y, Lee SH, Song I, Park JS, Cho YJ, Jo YH, Yoon HI, Lee JH, Lee CT, Lee YJ. Evaluation of the SpO2/FiO2 ratio as a predictor of intensive care unit transfers in respiratory ward patients for whom the rapid response system has been activated. PLoS One. 2018 Jul 31;13(7):e0201632. doi: 10.1371/journal.pone.0201632. eCollection 2018. PMID 30063769
- [Result] Wiedermann FJ, Stichlberger M, Glodny B. ARDS diagnosed by SpO2/FiO2 ratio compared with PaO2/FiO2 ratio: the role as a diagnostic tool for early enrolment into clinical trials. Open Med (Wars). 2016 Aug 2;11(1):297. doi: 10.1515/med-2016-0056. eCollection 2016. No abstract available. PMID 28352811
- [Derived] Kawaguchi A, Bernier G, Lacroix J, El Salti S, Cheng MP, Lee TC, Khwaja K, Jouvet P. Comparison of two methods to clear the airways of critically ill children and adults with COVID-19 infection: a structured summary of a study protocol for a pilot randomized controlled trial. Trials. 2020 Jul 3;21(1):610. doi: 10.1186/s13063-020-04533-6. PMID 32620174
- See also: Dymedso Inc. — https://www.dymedso.com/